CLINICAL TRIAL: NCT03411915
Title: A Phase 1 Multiple Dose Study to Evaluate the Safety and Tolerability of XmAb®18087 in Subjects With Advanced Neuroendocrine and Gastrointestinal Stromal Tumors (DUET-1)
Brief Title: A Study of XmAb®18087 in Subjects With NET and GIST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb18087-01; DUET-1 (Other: Xencor)
Record Dates: First submitted 2018-01-15; First posted 2018-01-26 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Neuroendocrine Tumor; Gastrointestinal Neoplasm
Keywords: NET; GIST; DUET-1
MeSH Terms: conditions — Neuroendocrine Tumors; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XmAb18087 (Experimental): XmAb18087 administered on days 1, 8, 15, and 22 of each 28-day cycle for a total of 3 cycles
  Interventions: Biological: XmAb18087

INTERVENTIONS:
Biological: XmAb18087 — monoclonal bispecific antibody

SUMMARY:
This is a Phase 1, multiple dose, ascending dose escalation study; to define a MTD/RD and regimen consisting of a first "priming" dose and escalated subsequent doses of XmAb18087; to describe safety and tolerability; to assess PK and immunogenicity; and to preliminarily assess anti-tumor activity of XmAb18087 in subjects with advanced NET or GIST.

The study will enroll dosing cohorts to establish a MTD/RD and regimen in subjects with advanced NET or GIST, then enroll additional subjects into separate NET and GIST expansion cohorts to collect additional data on safety and potential efficacy of XmAb18087.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed well differentiated low or intermediate grade (World Health Organization [WHO] Grade 1 or 2) NET of pancreatic, gastrointestinal, lung, or undetermined origin that is locally advanced or metastatic and has progressed within the past 12 months
* Histologically confirmed GIST that is locally advanced or metastatic
* NET and GIST tumors must be unresectable
* NET subjects must have progressed on or been ineligible for treatment with somatostatin analogues (SSA) and at least one other FDA-approved targeted therapy (everolimus or sunitinib).
* GIST subjects must have previously received all FDA-approved therapies (imatinib mesylate, sunitinib malate, and regorafenib) for which they are eligible
* Must have disease measurable by RECIST 1.1 criteria using either computed tomography (CT) or magnetic resonance imaging (MRI) scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Diagnosis of high-grade (WHO Grade 3) or poorly differentiated NET; high-grade neuroendocrine carcinoma; large cell neuroendocrine carcinoma, small cell carcinoma, or mixed small and large cell carcinoma.
* Subjects currently receiving anti-cancer therapies (other than SSAs, which may continue).
* Subjects who have received anti-cancer therapies within 2 weeks of the start of study drug (including chemotherapy, radiation therapy, immunotherapy, etc.).
* Must not be experiencing a Grade 3 or 4 toxicity from previous anti-cancer treatment
* Must not be receiving other anti-cancer therapies (except somatostatin analogues, which may be allowed)
* Must not have poorly controlled diabetes mellitus, known central nervous system involvement by malignant disease or insufficient bone marrow, renal, or hepatic function

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability profile of XmAb18087 | 84 Days
  Treatment-related adverse events as assessed by CTCAE v4.03
Identify the maximum tolerated dose (MTD) and/or recommended dose (RD) and schedule of XmAb18087 | 84 Days
  Establishing a safe and tolerable dose of XmAb18087 administered by intravenous (IV) dosing in NET and GIST patients

CONTACTS AND LOCATIONS:
Overall Officials: Zequn Tang, MD, PhD, Study Director — Senior Medical Director, Clinical Development, Xencor
Locations (16):
- United States (16):
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope Medical Center, Duarte, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - James Cancer Center, Columbus, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No